CLINICAL TRIAL: NCT07279337
Title: Effectiveness of Nutrition Counseling on Gestational Weight Gain Among Overweight and Obese Pregnant Women in Lebanon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nicosia (Other)
Responsible Party: Principal Investigator, Jessy Rizk, University instructor and dietitian, University of Nicosia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIUIRB-200706-JR1
Record Dates: First submitted 2025-11-30; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2021-02

CONDITIONS: Overweight and Obesity During Pregnancy
Keywords: Nutrition, pregnancy, obesity, dietary intervention, gestational weight gain
MeSH Terms: conditions — Overweight; Obesity; Gestational Weight Gain | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nutrition counseling provided by licensed dietitians (Experimental): The intervention group participated in an initial 30-60-minute nutrition counseling session with a registered dietitian during the first trimester.
  Counseling emphasized balanced nutrition, limiting added sugars and unhealthy fats, and promoting whole foods. Individualized weight gain targets were set based on Institute of Medicine (IOM) guidelines of 2009: 6.8-11.4 kg for overweight women and 5-9 kg for women with obesity. Participants were also advised to engage in 150 minutes of moderate-intensity physical activity per week, as recommended by health guidelines.
  Follow-ups were conducted every 10-15 days via smartphone applications (e.g., WhatsApp, Zoom) with an average of 14 nutrition follow-ups throughout the intervention. The follow-ups were utilizing asynchronous telehealth platform that was secure and user-friendly.
  Interventions: Behavioral: Intervention group that received detailed nutrition assessment, counseling, and monitoring
- Control group (No Intervention): Usual prenatal care

INTERVENTIONS:
Behavioral: Intervention group that received detailed nutrition assessment, counseling, and monitoring — The intervention group participated in an initial 30-60-minute nutrition counseling session with a registered dietitian during the first trimester.
  Counseling emphasized balanced nutrition, limiting added sugars and unhealthy fats, and promoting whole foods. Individualized weight gain targets were set based on Institute of Medicine (IOM) guidelines of 2009: 6.8-11.4 kg for overweight women and 5-9 kg for women with obesity. Participants were also advised to engage in 150 minutes of moderate-intensity physical activity per week, as recommended by health guidelines.
  Follow-ups were conducted every 10-15 days via smartphone applications (e.g., WhatsApp, Zoom) with an average of 14 nutrition follow-ups throughout the intervention. The follow-ups were utilizing asynchronous telehealth platform that was secure
  Arms: nutrition counseling provided by licensed dietitians

SUMMARY:
A high percentage of women are either overweight or obese before pregnancy and many women are exceeding the gestational weight gain recommendations when pregnant. Excessive gestational weight gain increases the risk of maternal and fetal complications. To help with this, women need to be advised about the appropriate weight gain recommendation according to their pre-pregnancy body weight. One way to do this is by receiving dietary and lifestyle advices during prenatal visits. This study will contribute to knowledge that will inform dietary guidelines and public policy on how to manage gestational weight gain and thus improve maternal and fetal outcomes.

DETAILED DESCRIPTION:
If you choose to participate in the suggested study, you will be seen by a dietitian during the first trimester for an in-depth counseling session and provide you with individualized nutrition counseling regarding your physical activity, dietary, and weight gain goals. You will then be asked to self-monitor your diet, weight, and physical activity. Study staff will instruct you on how to keep weekly paper logs of weight, activity, and diet that you will share with your dietitian weekly or biweekly by telephone. In order to determine the total gestational weight gain and to determine the impact of nutrition intervention on the health of your baby, data collectors will review your medical record to obtain your weight at delivery, your infants' birthweight, and method of delivery.

Apart from the 30 minutes of your time taken during the nutrition counseling session and your dietary and activity commitment according to the recommendations, we can expect no risks or inconveniences for you. Your participation in the study is voluntary and you may withdraw your participation from the study at any time. Your personal health information will be treated as confidential and all persons involved in the study are committed to respecting your privacy.

ELIGIBILITY:
Inclusion Criteria:

* In their first trimester of pregnancy
* With a pre-pregnancy Body Mass Index (BMI) ranging from 25 to 35 kg/m², classifying them as overweight or obese.
* Women were required to be attending regular prenatal care visits at randomly selected gynecology clinics

  * The ability and willingness to meet with a licensed dietitian for individualized counseling.
  * Commitment to follow the recommended nutrition and physical activity guidelines throughout the duration of the study

Exclusion Criteria:

* Contraindications to exercise
* Medical conditions such as uncontrolled hypertension, insulin-dependent diabetes, uncontrolled thyroid disease, multiple gestation, persistent bleeding in the first trimester
* History of recurrent miscarriages.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | 6-8 months period
  Total weight gained during pregnancy

SECONDARY OUTCOMES:
adherence to IOM weight gain guidelines | 1 month
  comparing actual gestational weight gain to guidelines based on pre-BMI category

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese International University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided
It depends on what information is needed. Values like gestational weight gain of participants can be shared.